CLINICAL TRIAL: NCT02074254
Title: Safety of Percutaneous Tracheostomy in Clopidogrel and Selective Serotonin Reuptake Inhibitors
Status: Withdrawn | Type: Observational
Why Stopped: Not sure. PI is no longer at OSU.
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012E0196
Record Dates: First submitted 2013-06-04; First posted 2014-02-28 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Tracheostomy Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Safety of Percutaneous Tracheostomy in Clopidogrel and Selective Serotonin Reuptake Inhibitors

DETAILED DESCRIPTION:
We propose a retrospective review of our experience with bleeding complication in the presence of antiplatelet and SSRI therapy and compare the complications with those who were not on antiplatelet agents or SSRI.

ELIGIBILITY:
Inclusion Criteria:

* on antiplatelet therapy or selective serotonin reuptake inhibitors(SSRI)

Exclusion Criteria:

* N/A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is being done to evaluate the safety of percutaneous tracheostomy in patients taking antiplatelet agents such as aspirin and/ or clopidogrel or selective serotonin reuptake inhibitors. We will identify all patients age 18 or older who have undergone percutaneous tracheostomy by interventional pulmonology at OSUMC and access their PHI to record variables (see data collection form).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03-22 (Actual); Primary Completion 2012-05-09 (Estimated); Study Completion 2012-05-09 (Estimated)

PRIMARY OUTCOMES:
a retrospective review of our experience with bleeding complication in the presence of antiplatelet and SSRI therapy and compare the complications with those who were not on antiplatelet agents or SSRI | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Islam, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - OSUMC, Columbus, Ohio
  - University Hospital, OSUMC 473 W 12th Ave, Columbus, Ohio